CLINICAL TRIAL: NCT02098590
Title: Chemoprophylaxis and Plasmodium Falciparum NF54 Sporozoite Immunization Challenged by Heterologous Infection
Acronym: BMGF2b
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BMGF2b
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Malaria
Keywords: Malaria; Plasmodium falciparum
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — atovaquone, proguanil drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- NF54 CPS-immunization challenged by NF135.C10 (Experimental): Subjects will receive CPS-immunization by bites from 3 x 15 NF54 P. falciparum infected mosquitoes under chloroquine prophylaxis. After stopping chloroquine subjects will receive a heterologous malaria challenge infection by exposure to the bites of 5 NF135.C10 P. falciparum infected mosquitoes. Subjects will be treated with Malarone if they develop a malaria infection or on day 28 after challenge infection.
  Interventions: Biological: CPS-immunization; Biological: malaria challenge infection, P. falciparum NF135.C10; Drug: atovaquone/proguanil
- NF54 CPS-immunization challenged by NF166.C8 (Experimental): Subjects will receive CPS-immunization by bites from 3 x 15 NF54 P. falciparum infected mosquitoes under chloroquine prophylaxis. After stopping chloroquine subjects will receive a heterologous malaria challenge infection by exposure to the bites of 5 NF166.C8 P. falciparum infected mosquitoes. Subjects will be treated with Malarone if they develop a malaria infection or on day 28 after challenge infection.
  Interventions: Biological: CPS-immunization; Biological: malaria challenge infection, P. falciparum NF166.C8; Drug: atovaquone/proguanil
- NF54 CPS-immunization challenged by NF54 (Other): [Negative control group, to assess effectiveness of CPS-immunization.] Subjects will receive CPS-immunization by bites from 3 x 15 NF54 P. falciparum infected mosquitoes under chloroquine prophylaxis. After stopping chloroquine subjects will receive a homologous malaria challenge infection by exposure to the bites of 5 NF54 P. falciparum infected mosquitoes. Subjects will be treated with Malarone if they develop a malaria infection or on day 28 after challenge infection.
  Interventions: Biological: CPS-immunization; Biological: malaria challenge infection, P. falciparum NF54; Drug: atovaquone/proguanil
- Control group challenged by NF135.C10 (Other): [Control group] Subjects will receive bites from 3 x 15 uninfected mosquitoes under chloroquine prophylaxis. After stopping chloroquine subjects will receive a malaria challenge infection by exposure to the bites of NF135.C10 P. falciparum infected mosquitoes. Subjects will be treated with Malarone if they develop a malaria infection or on day 28 after challenge infection.
  Interventions: Biological: malaria challenge infection, P. falciparum NF135.C10; Drug: atovaquone/proguanil
- Control group challenged by NF166.C8 (Other): [Control group] Subjects will receive bites from 3 x 15 uninfected mosquitoes under chloroquine prophylaxis. After stopping chloroquine subjects will receive a malaria challenge infection by exposure to the bites of NF166.C8 P. falciparum infected mosquitoes. Subjects will be treated with Malarone if they develop a malaria infection or on day 28 after challenge infection.
  Interventions: Biological: malaria challenge infection, P. falciparum NF166.C8; Drug: atovaquone/proguanil
- Control group challenged by NF54 (Other): [Control group] Subjects will receive bites from 3 x 15 uninfected mosquitoes under chloroquine prophylaxis. After stopping chloroquine subjects will receive a malaria challenge infection by exposure to the bites of NF54 P. falciparum infected mosquitoes. Subjects will be treated with Malarone if they develop a malaria infection or on day 28 after challenge infection.
  Interventions: Biological: malaria challenge infection, P. falciparum NF54; Drug: atovaquone/proguanil

INTERVENTIONS:
Biological: CPS-immunization — Subjects will be exposed 3 times to bites from 15 NF54 Plasmodium infected mosquitoes during each immunization, while taking chloroquin prophylaxis.
  Other Names: chloroquin; Plasmodium falciparum NF54 sporozoites
  Arms: NF54 CPS-immunization challenged by NF135.C10; NF54 CPS-immunization challenged by NF166.C8; NF54 CPS-immunization challenged by NF54
Biological: malaria challenge infection, P. falciparum NF135.C10 — Subjects will receive bites from 5 Anopheles mosquitoes infected with Plasmodium falciparum NF135.C10 sporozoites.
  Other Names: Plasmodium falciparum NF135.C10 sporozoites
  Arms: Control group challenged by NF135.C10; NF54 CPS-immunization challenged by NF135.C10
Biological: malaria challenge infection, P. falciparum NF166.C8 — Subjects will receive bites from 5 Anopheles mosquitoes infected with Plasmodium falciparum NF166.C8 sporozoites.
  Other Names: Plasmodium falciparum NF166.C8 sporozoites
  Arms: Control group challenged by NF166.C8; NF54 CPS-immunization challenged by NF166.C8
Biological: malaria challenge infection, P. falciparum NF54 — Subjects will receive bites from 5 Anopheles mosquitoes infected with Plasmodium falciparum NF54 sporozoites.
  Other Names: Plasmodium falciparum NF54 sporozoites
  Arms: Control group challenged by NF54; NF54 CPS-immunization challenged by NF54
Drug: atovaquone/proguanil — All participants will be treated with atovaquone/proguanil when they develop a malaria infection or on day 28 after malaria challenge infection.
  Other Names: Malarone

SUMMARY:
Malaria, a disease caused by the parasite Plasmodium, is one of the world's major infectious diseases. With approximately 627.000 deaths a year, it is both a chief cause of morbidity and mortality as well as a significant contribution to ongoing poverty in endemic countries. Ultimately, the key to malaria control, and hopefully eradication, would be an effective vaccine. Though a number of vaccine-candidates have entered the pipeline of pre-clinical and clinical development, they have yet to achieve the level of efficacy necessary for effective malaria prevention. It has been shown previously that if healthy human volunteers taking chloroquine chemoprophylaxis are repeatedly exposed to Plasmodium parasites through the bites of infected mosquitoes, they are fully protected against a later challenge infection with a 'homologous' (genetically similar) Plasmodium parasite. This process is known as ChemoProphylaxis and Sporozoites, or CPS-immunization. One of the obstacles to developing an effective vaccine is the genetic heterogeneity of malaria parasites. To further consider the development of whole-parasite based vaccines against malaria and in order to better understand the protective immunity induced by CPS-immunization, it is essential to investigate whether heterologous protection against genetically diverse (heterologous) P. falciparum clones can be induced.

This is a single center, randomized, double-blind study to determine whether healthy volunteers immunized with P. falciparum NF54 parasites under chloroquine prophylaxis are protected against a challenge infection with the genetically distinct NF135.C10 or NF166.C8 P. falciparum clones.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. Subject is aged ≥ 18 and ≤ 35 years and in good health.
2. Subject has adequate understanding of the procedures of the study and agrees to abide strictly thereby.
3. Subject is able to communicate well with the investigator, is available to attend all study visits, lives in proximity to the trial centre (<10 km) or (if >10km) is willing to stay in a hotel close to the trial centre during part of the study (day 5 post-infection until three days post-treatment). Furthermore the subject will remain within the Netherlands during the challenge period, not travel to a malaria-endemic area during the study period, and is reachable (24/7) by mobile telephone throughout the entire study period.
4. Subject agrees to inform his/her general practitioner about participation in the study and to sign a request to release by the General Practitioner (GP) any relevant medical information concerning possible contra-indications for participation in the study.
5. Subject agrees to refrain from blood donation to Sanquin or for other purposes throughout the study period and for a defined period thereafter according to current Sanquin guidelines.
6. For female subjects: subject agrees to use adequate contraception and not to breastfeed for the duration of study.
7. Subject has signed informed consent.
8. Subject agrees to refrain from intensive physical exercise (disproportionate to the subjects usual daily activity or exercise routine) for ten days following each immunization and during the malaria challenge period.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, renal, hepatic, neurological, dermatological, endocrine, malignant, haematological, infectious, immunodeficient, psychiatric and other disorders, which could compromise the health of the volunteer during the study or interfere with the interpretation of the study results. These include, but are not limited to, any of the following.

   1.1 Body weight <50 kg or Body Mass Index (BMI) <18.0 or >30.0 kg/m2 at screening.

   1.2 A heightened risk of cardiovascular disease, as determined by: an estimated ten year risk of fatal cardiovascular disease of ≥5% at screening, as determined by the Systematic Coronary Risk Evaluation (SCORE); history, or evidence at screening, of clinically significant arrhythmia's, prolonged QT-interval or other clinically relevant ECG abnormalities; or a positive family history of cardiac events in 1st or 2nd degree relatives <50 years old.

   1.3 A medical history of functional asplenia, sickle cell trait/disease, thalassaemia trait/disease or G6PD deficiency.

   1.4 History of epilepsy in the period of five years prior to study onset, even if no longer on medication.

   1.5 Positive Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) screening tests.

   1.6 Chronic use of i) immunosuppressive drugs, ii) antibiotics, iii) or other immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period.

   1.7 History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years.

   1.8 Any history of treatment for severe psychiatric disease by a psychiatrist in the past year.

   1.9 History of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset, positive urine toxicology test for cocaine or amphetamines at screening or prior to infection or positive urine toxicology test for cannabis at inclusion or prior to infection.
2. For female subjects: positive urine pregnancy test at screening or prior to infection.
3. Any history of malaria, positive serology for P. falciparum, or previous participation in any malaria (vaccine) study.
4. Known hypersensitivity to or contra-indications (including co-medication) for use of chloroquine, Malarone or artemether-lumefantrine, or history of severe (allergic) reactions to mosquito bites.
5. Receipt of any vaccinations in the 3 months prior to the start of the study or plans to receive any other vaccinations during the study period or up to 8 weeks thereafter.
6. Participation in any other clinical study in the 30 days prior to the start of the study or during the study period.
7. Being an employee or student of the department of Medical Microbiology of the Radboudumc or the department of Internal Medicine.
8. Any other condition or situation that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Parasitemia | day 1 - 28 after malaria challenge infection
  The effectiveness of CPS-immunization with NF54 sporozoites to protect against malaria challenge infection with heterologous NF135.C10 or NF166.C8 sporozoites will be determined by the time to parasitemia in immunized versus non-immunized volunteers after the challenge infection.

SECONDARY OUTCOMES:
Antigen specificity of CPS-immunization induced antibodies against P. falciparum | 6-10 days after challenge infection
  Blood will be drawn to isolate plasmablast for further delineation of the antibody responses following CPS-immunization.
Specificity of CPS-immunization induced T-cell responses against P. falciparum | 14 days after each CPS-immunization
  Blood will be drawn to isolate monocytes and T cells, which will be used to determine the activity of T cells against specific target antigens of the pre-erythrocytic stages of Plasmodium falciparum.

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Sauerwein, Prof, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Roestenberg M, McCall M, Hopman J, Wiersma J, Luty AJ, van Gemert GJ, van de Vegte-Bolmer M, van Schaijk B, Teelen K, Arens T, Spaarman L, de Mast Q, Roeffen W, Snounou G, Renia L, van der Ven A, Hermsen CC, Sauerwein R. Protection against a malaria challenge by sporozoite inoculation. N Engl J Med. 2009 Jul 30;361(5):468-77. doi: 10.1056/NEJMoa0805832. PMID 19641203
- [Background] Roestenberg M, O'Hara GA, Duncan CJ, Epstein JE, Edwards NJ, Scholzen A, van der Ven AJ, Hermsen CC, Hill AV, Sauerwein RW. Comparison of clinical and parasitological data from controlled human malaria infection trials. PLoS One. 2012;7(6):e38434. doi: 10.1371/journal.pone.0038434. Epub 2012 Jun 11. PMID 22701640
- [Derived] Walk J, Reuling IJ, Behet MC, Meerstein-Kessel L, Graumans W, van Gemert GJ, Siebelink-Stoter R, van de Vegte-Bolmer M, Janssen T, Teelen K, de Wilt JHW, de Mast Q, van der Ven AJ, Diez Benavente E, Campino S, Clark TG, Huynen MA, Hermsen CC, Bijker EM, Scholzen A, Sauerwein RW. Modest heterologous protection after Plasmodium falciparum sporozoite immunization: a double-blind randomized controlled clinical trial. BMC Med. 2017 Sep 13;15(1):168. doi: 10.1186/s12916-017-0923-4. PMID 28903777